CLINICAL TRIAL: NCT01459705
Title: Comparing Virtual Reality Exposure Therapy to Prolonged Exposure in the Treatment of Soldiers With Post Traumatic Stress Disorder (PTSD)
Brief Title: Comparing Virtual Reality Exposure Therapy to Prolonged Exposure
Acronym: VRPE Extension
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Center for Telehealth and Technology (U.S. Federal Agency)
Collaborators: The Geneva Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 112226; W81XWH-11-2-0007 (Other Grant/Funding Number: USMRMC)
Record Dates: First submitted 2011-10-24; First posted 2011-10-26 (Estimated); Results first posted 2015-12-14 (Estimated); Last update posted 2015-12-14 (Estimated); Status verified 2015-11

CONDITIONS: Stress Disorders; Post-Traumatic Stress Disorder
Keywords: Combat Disorders; Exposure Therapy; Army Personnel
MeSH Terms: conditions — Stress Disorders, Traumatic; Stress Disorders, Post-Traumatic; Combat Disorders | interventions — Virtual Reality Exposure Therapy; Waiting Lists

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Prolonged Exposure Therapy (PE) (Active Comparator): The PE protocol is based on manualized procedures, which are derived from the theory that effective treatment for PTSD requires that the underlying pathological fear structure be activated and paired with new information that is incompatible with the fear structure. PE involves imaginal exposure and in vivo exposure as the two primary strategies to elicit repeated confrontation of feared but objectively safe thoughts, feelings, situations and events.
  Interventions: Behavioral: Prolonged Exposure Therapy (PE)
- Virtual Reality Exposure Therapy (VRET) (Experimental): The VRET protocol follows the same procedures as the PE protocol with the primary exception being that all instances of imaginal exposure will be augmented by immersion into Virtual Iraq environments, thus creating a situation known as immersive exposure.
  Interventions: Behavioral: Virtual Reality Exposure Therapy (VRET)
- Waitlist (Placebo Comparator): The waitlist (WL) participants will be asked to refrain from psychotherapy during the 5 weeks of study participation.
  Interventions: Behavioral: Waitlist

INTERVENTIONS:
Behavioral: Prolonged Exposure Therapy (PE) — Prolonged exposure therapy will consist of 10 treatment sessions lasting 90 - 120 minutes each, with additional between-session homework assignments.
  Other Names: PE
  Arms: Prolonged Exposure Therapy (PE)
Behavioral: Virtual Reality Exposure Therapy (VRET) — Virtual Reality Exposure Therapy will consist of 10 treatment sessions lasting 90 -120 minutes with additional between-session homework assignments.
  Other Names: VRE; VRET
  Arms: Virtual Reality Exposure Therapy (VRET)
Behavioral: Waitlist — This group will refrain from psychotherapy until after the completion of the 5 weeks of study participation
  Other Names: WL; Waitlist Control Group
  Arms: Waitlist

SUMMARY:
This study is evaluating the efficacy of virtual reality exposure therapy (VRET) by comparing it to prolonged exposure therapy (PE) and a waitlist(WL) group for the treatment of post traumatic stress disorder (PTSD) in active duty (AD) Soldiers with combat-related trauma. The investigators will test the general hypothesis that 10 sessions of VRET or PE will successfully treat PTSD, therapeutically affect levels of physiological arousal, and significantly reduce perceptions of stigma toward seeking behavioral health services.

DETAILED DESCRIPTION:
The rationale for this study is based on growing evidence demonstrating that VRET is an efficacious treatment for PTSD and holds the potential to improve access to care for Soldiers who would otherwise avoid treatment. Although PE is considered one of the most effective cognitive-behavioral therapies (CBT) for treatments for PTSD, there are reasons why it may not be the most viable option for many Soldiers. First, prolonged exposure requires a level of emotional engagement during exposure to the trauma that many patients are unable to obtain. Second, stigma and concerns about how Soldiers will be perceived by peers and leadership has a dramatic impact on whether a Soldier will seek care. VRET may address these concerns and may also improve treatment outcomes and access to care by augmenting the patient's re-living of the trauma with a sensory-rich environment and moderating stigma perceptions by offering non-traditional treatment that is a preferable option for many Soldiers who are reluctant to seek out traditional talk therapies. Despite its promise as a viable treatment option, few studies have examined VRET for combat-related PTSD and there are no published studies that have compared VRET to PE in the treatment of combat-related PTSD. Positive results may provide new treatment options for all Soldiers, but should prove to be an especially attractive option for Soldiers who either do not respond to, or are reluctant to engage in other established therapies such as PE.

ELIGIBILITY:
Inclusion Criteria:

* PTSD diagnosis as assessed by CAPS
* history of deployment in support of Operation Iraqi Freedom/ Operation Enduring Freedom(OIF/OEF)
* non sexually based deployment related trauma
* three or more months since index trauma
* stable on psychotropic medication for 30 days

Exclusion Criteria:

* index trauma in the last three months
* history of schizophrenia, other psychotic or bipolar disorder
* history of organic brain disorder
* suicidal risk or intent or self-mutilating behavior requiring hospitalization in the last 6 months
* ongoing threatening situation
* current drug or alcohol dependence
* history of seizures
* prior history of PE for PTSD
* other current psychotherapy
* physical condition that interferes with proper use of Virtual Reality head mounted display
* history of loss of consciousness since entering active duty service greater than 15 minutes history of schizophrenia, other psychotic or bipolar disorder

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 162 (Actual)
Dates: Start 2011-10; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gregory A Gahm, PhD, Principal Investigator — DCoE- National Center for Telehealth and Technology; Greg Reger, PhD, Principal Investigator — DCoE - National Center for Telehealth and Technology
Locations (1):
- Womack Clinical Psychology Service, Fort Bragg, North Carolina, United States

REFERENCES:
- [Background] Difede J, Cukor J, Patt I, Giosan C, Hoffman H. The application of virtual reality to the treatment of PTSD following the WTC attack. Ann N Y Acad Sci. 2006 Jul;1071:500-1. doi: 10.1196/annals.1364.052. PMID 16891607
- [Background] Rothbaum BO, Hodges LF, Ready D, Graap K, Alarcon RD. Virtual reality exposure therapy for Vietnam veterans with posttraumatic stress disorder. J Clin Psychiatry. 2001 Aug;62(8):617-22. doi: 10.4088/jcp.v62n0808. PMID 11561934
- [Background] Koenen KC, Stellman JM, Stellman SD, Sommer JF Jr. Risk factors for course of posttraumatic stress disorder among Vietnam veterans: a 14-year follow-up of American Legionnaires. J Consult Clin Psychol. 2003 Dec;71(6):980-6. doi: 10.1037/0022-006X.71.6.980. PMID 14622073
- [Background] Bryant RA, Moulds ML, Guthrie RM, Dang ST, Nixon RD. Imaginal exposure alone and imaginal exposure with cognitive restructuring in treatment of posttraumatic stress disorder. J Consult Clin Psychol. 2003 Aug;71(4):706-12. doi: 10.1037/0022-006x.71.4.706. PMID 12924676
- [Background] Foa EB. Psychosocial treatment of posttraumatic stress disorder. J Clin Psychiatry. 2000;61 Suppl 5:43-8; discussion 49-51. PMID 10761678
- [Background] Foa EB, Meadows EA. Psychosocial treatments for posttraumatic stress disorder: a critical review. Annu Rev Psychol. 1997;48:449-80. doi: 10.1146/annurev.psych.48.1.449. PMID 9046566
- [Background] Carlson JG, Chemtob CM, Rusnak K, Hedlund NL, Muraoka MY. Eye movement desensitization and reprocessing (EDMR) treatment for combat-related posttraumatic stress disorder. J Trauma Stress. 1998 Jan;11(1):3-24. doi: 10.1023/A:1024448814268. PMID 9479673
- [Background] Sherman JJ. Effects of psychotherapeutic treatments for PTSD: a meta-analysis of controlled clinical trials. J Trauma Stress. 1998 Jul;11(3):413-35. doi: 10.1023/A:1024444410595. PMID 9690185
- [Background] Bisson J, Andrew M. Psychological treatment of post-traumatic stress disorder (PTSD). Cochrane Database Syst Rev. 2005 Apr 18;(2):CD003388. doi: 10.1002/14651858.CD003388.pub2. PMID 15846661
- [Background] Resick PA, Nishith P, Weaver TL, Astin MC, Feuer CA. A comparison of cognitive-processing therapy with prolonged exposure and a waiting condition for the treatment of chronic posttraumatic stress disorder in female rape victims. J Consult Clin Psychol. 2002 Aug;70(4):867-79. doi: 10.1037//0022-006x.70.4.867. PMID 12182270
- [Background] Foa EB, Kozak MJ. Emotional processing of fear: exposure to corrective information. Psychol Bull. 1986 Jan;99(1):20-35. No abstract available. PMID 2871574
- [Background] Delahanty DL, Raimonde AJ, Spoonster E. Initial posttraumatic urinary cortisol levels predict subsequent PTSD symptoms in motor vehicle accident victims. Biol Psychiatry. 2000 Nov 1;48(9):940-7. doi: 10.1016/s0006-3223(00)00896-9. PMID 11074232
- [Background] Shalev AY, Sahar T, Freedman S, Peri T, Glick N, Brandes D, Orr SP, Pitman RK. A prospective study of heart rate response following trauma and the subsequent development of posttraumatic stress disorder. Arch Gen Psychiatry. 1998 Jun;55(6):553-9. doi: 10.1001/archpsyc.55.6.553. PMID 9633675
- [Background] Mason J, Southwick S, Yehuda R, Wang S, Riney S, Bremner D, Johnson D, Lubin H, Blake D, Zhou G, et al. Elevation of serum free triiodothyronine, total triiodothyronine, thyroxine-binding globulin, and total thyroxine levels in combat-related posttraumatic stress disorder. Arch Gen Psychiatry. 1994 Aug;51(8):629-41. doi: 10.1001/archpsyc.1994.03950080041006. PMID 8042912
- [Background] Yehuda R. Post-traumatic stress disorder. N Engl J Med. 2002 Jan 10;346(2):108-14. doi: 10.1056/NEJMra012941. No abstract available. PMID 11784878
- [Background] Yehuda R, Siever LJ, Teicher MH, Levengood RA, Gerber DK, Schmeidler J, Yang RK. Plasma norepinephrine and 3-methoxy-4-hydroxyphenylglycol concentrations and severity of depression in combat posttraumatic stress disorder and major depressive disorder. Biol Psychiatry. 1998 Jul 1;44(1):56-63. doi: 10.1016/s0006-3223(98)80007-3. PMID 9646884
- [Background] Morgan CA 3rd, Grillon C, Southwick SM, Davis M, Charney DS. Exaggerated acoustic startle reflex in Gulf War veterans with posttraumatic stress disorder. Am J Psychiatry. 1996 Jan;153(1):64-8. doi: 10.1176/ajp.153.1.64. PMID 8540594
- [Background] Shalev AY, Peri T, Orr SP, Bonne O, Pitman RK. Auditory startle responses in help-seeking trauma survivors. Psychiatry Res. 1997 Mar 3;69(1):1-7. doi: 10.1016/s0165-1781(96)03001-6. PMID 9080539
- [Background] Malloy PF, Fairbank JA, Keane TM. Validation of a multimethod assessment of posttraumatic stress disorders in Vietnam veterans. J Consult Clin Psychol. 1983 Aug;51(4):488-94. doi: 10.1037//0022-006x.51.4.488. No abstract available. PMID 6619355
- [Background] Orr SP, Lasko NB, Shalev AY, Pitman RK. Physiologic responses to loud tones in Vietnam veterans with posttraumatic stress disorder. J Abnorm Psychol. 1995 Feb;104(1):75-82. doi: 10.1037//0021-843x.104.1.75. PMID 7897056
- [Background] Pitman RK, Orr SP, Altman B, Longpre RE, Poire RE, Macklin ML, Michaels MJ, Steketee GS. Emotional processing and outcome of imaginal flooding therapy in Vietnam veterans with chronic posttraumatic stress disorder. Compr Psychiatry. 1996 Nov-Dec;37(6):409-18. doi: 10.1016/s0010-440x(96)90024-3. PMID 8932965
- [Background] Keane TM, Kaloupek DG. Imaginal flooding in the treatment of a posttraumatic stress disorder. J Consult Clin Psychol. 1982 Feb;50(1):138-40. doi: 10.1037//0022-006x.50.1.138. No abstract available. PMID 7056906
- [Background] Cardena E, Spiegel D. Dissociative reactions to the San Francisco Bay Area earthquake of 1989. Am J Psychiatry. 1993 Mar;150(3):474-8. doi: 10.1176/ajp.150.3.474. PMID 8434665
- [Background] Koopman C, Classen C, Spiegel D. Predictors of posttraumatic stress symptoms among survivors of the Oakland/Berkeley, Calif., firestorm. Am J Psychiatry. 1994 Jun;151(6):888-94. doi: 10.1176/ajp.151.6.888. PMID 8184999
- [Background] Reger GM, McGee JS, van der Zaag C, Thiebaux M, Galen Buckwalter JG, Rizzo AA. A 3D virtual environment rod and frame test: the reliability and validity of four traditional scoring methods for older adults. J Clin Exp Neuropsychol. 2003 Dec;25(8):1169-77. doi: 10.1076/jcen.25.8.1169.16733. PMID 14566588
- [Background] Rothbaum BO, Hodges L, Watson BA, Kessler CD, Opdyke D. Virtual reality exposure therapy in the treatment of fear of flying: a case report. Behav Res Ther. 1996 May-Jun;34(5-6):477-81. doi: 10.1016/0005-7967(96)00007-1. PMID 8687369
- [Background] Rothbaum BO, Hodges L, Smith S, Lee JH, Price L. A controlled study of virtual reality exposure therapy for the fear of flying. J Consult Clin Psychol. 2000 Dec;68(6):1020-6. doi: 10.1037//0022-006x.68.6.1020. PMID 11142535
- [Background] Rothbaum BO, Hodges L, Anderson PL, Price L, Smith S. Twelve-month follow-up of virtual reality and standard exposure therapies for the fear of flying. J Consult Clin Psychol. 2002 Apr;70(2):428-32. doi: 10.1037//0022-006x.70.2.428. PMID 11952201
- [Background] Rothbaum BO, Hodges LF, Kooper R, Opdyke D, Williford JS, North M. Effectiveness of computer-generated (virtual reality) graded exposure in the treatment of acrophobia. Am J Psychiatry. 1995 Apr;152(4):626-8. doi: 10.1176/ajp.152.4.626. PMID 7694917
- [Background] Emmelkamp PM, Krijn M, Hulsbosch AM, de Vries S, Schuemie MJ, van der Mast CA. Virtual reality treatment versus exposure in vivo: a comparative evaluation in acrophobia. Behav Res Ther. 2002 May;40(5):509-16. doi: 10.1016/s0005-7967(01)00023-7. PMID 12038644
- [Background] Botella C, Banos RM, Perpina C, Villa H, Alcaniz M, Rey A. Virtual reality treatment of claustrophobia: a case report. Behav Res Ther. 1998 Feb;36(2):239-46. doi: 10.1016/s0005-7967(97)10006-7. PMID 9613029
- [Background] Carlin AS, Hoffman HG, Weghorst S. Virtual reality and tactile augmentation in the treatment of spider phobia: a case report. Behav Res Ther. 1997 Feb;35(2):153-8. doi: 10.1016/s0005-7967(96)00085-x. PMID 9046678
- [Background] Garcia-Palacios A, Hoffman H, Carlin A, Furness TA 3rd, Botella C. Virtual reality in the treatment of spider phobia: a controlled study. Behav Res Ther. 2002 Sep;40(9):983-93. doi: 10.1016/s0005-7967(01)00068-7. PMID 12296495
- [Background] Rothbaum BO, Anderson P, Zimand E, Hodges L, Lang D, Wilson J. Virtual reality exposure therapy and standard (in vivo) exposure therapy in the treatment of fear of flying. Behav Ther. 2006 Mar;37(1):80-90. doi: 10.1016/j.beth.2005.04.004. Epub 2006 Feb 24. PMID 16942963
- [Background] Botella C, Perpina C, Banos RM, Garcia-Palacios A. Virtual reality: a new clinical setting lab. Stud Health Technol Inform. 1998;58:73-81. PMID 10350931
- [Background] Gershon J, Zimand E, Lemos R, Rothbaum BO, Hodges L. Use of virtual reality as a distractor for painful procedures in a patient with pediatric cancer: a case study. Cyberpsychol Behav. 2003 Dec;6(6):657-61. doi: 10.1089/109493103322725450. PMID 14756933
- [Background] Rothbaum BO, Hodges L, Alarcon R, Ready D, Shahar F, Graap K, Pair J, Hebert P, Gotz D, Wills B, Baltzell D. Virtual reality exposure therapy for PTSD Vietnam Veterans: a case study. J Trauma Stress. 1999 Apr;12(2):263-71. doi: 10.1023/A:1024772308758. PMID 10378165
- [Background] Bradley R, Greene J, Russ E, Dutra L, Westen D. A multidimensional meta-analysis of psychotherapy for PTSD. Am J Psychiatry. 2005 Feb;162(2):214-27. doi: 10.1176/appi.ajp.162.2.214. PMID 15677582
- [Background] Blake DD, Weathers FW, Nagy LM, Kaloupek DG, Gusman FD, Charney DS, Keane TM. The development of a Clinician-Administered PTSD Scale. J Trauma Stress. 1995 Jan;8(1):75-90. doi: 10.1007/BF02105408. PMID 7712061
- [Background] Aziz MA, Kenford S. Comparability of telephone and face-to-face interviews in assessing patients with posttraumatic stress disorder. J Psychiatr Pract. 2004 Sep;10(5):307-13. doi: 10.1097/00131746-200409000-00004. PMID 15361745
- [Background] Blanchard EB, Jones-Alexander J, Buckley TC, Forneris CA. Psychometric properties of the PTSD Checklist (PCL). Behav Res Ther. 1996 Aug;34(8):669-73. doi: 10.1016/0005-7967(96)00033-2. PMID 8870294
- [Background] Bolton EE, Gray MJ, Litz BT. A cross-lagged analysis of the relationship between symptoms of PTSD and retrospective reports of exposure. J Anxiety Disord. 2006;20(7):877-95. doi: 10.1016/j.janxdis.2006.01.009. Epub 2006 Mar 10. PMID 16530379
- [Background] Beck AT, Steer RA, Ball R, Ranieri W. Comparison of Beck Depression Inventories -IA and -II in psychiatric outpatients. J Pers Assess. 1996 Dec;67(3):588-97. doi: 10.1207/s15327752jpa6703_13. PMID 8991972
- [Background] Beck AT, Epstein N, Brown G, Steer RA. An inventory for measuring clinical anxiety: psychometric properties. J Consult Clin Psychol. 1988 Dec;56(6):893-7. doi: 10.1037//0022-006x.56.6.893. No abstract available. PMID 3204199
- [Background] Mackenzie CS, Gekoski WL, Knox VJ. Age, gender, and the underutilization of mental health services: the influence of help-seeking attitudes. Aging Ment Health. 2006 Nov;10(6):574-82. doi: 10.1080/13607860600641200. PMID 17050086
- [Background] Pyne JM, Kuc EJ, Schroeder PJ, Fortney JC, Edlund M, Sullivan G. Relationship between perceived stigma and depression severity. J Nerv Ment Dis. 2004 Apr;192(4):278-83. doi: 10.1097/01.nmd.0000120886.39886.a3. PMID 15060401
- [Background] Larsen DL, Attkisson CC, Hargreaves WA, Nguyen TD. Assessment of client/patient satisfaction: development of a general scale. Eval Program Plann. 1979;2(3):197-207. doi: 10.1016/0149-7189(79)90094-6. No abstract available. PMID 10245370
- [Background] Bryant RA. Cognitive behavior therapy of violence-related posttraumatic stress disorder. Aggression and Violent Behavior. 2000;5:79-97.
- [Background] Foa EB,Steketee GS, Rothbaum BO. Behavioral/cognitive conceptualizations of post-traumatic stress disorder. Behavior Therapy. 1989;20:155-176.
- [Background] Foa EB, Hearst-Ikeda D. Emotional Dissociation in Response to Trauma: An Information-Processing Approach. In: Michelson LK, Ray WJ, eds. Handbook of Dissociation: Theoretical and Clinical Perspectives. New York: Plenum Press; 1996:207-222.
- [Background] Lating JM, Everly GS, Jr. Psychophysiological assessment of PTSD. In: Everly, GS, Jr., Lating LM, eds. Psychotraumatology: Key papers and core concepts in post-traumatic stress. New York: Plenum Press; 1995:129-145.
- [Background] Boudewyns P, Hyer L. Physiological response to combat memories and preliminary treatment outcome in Vietnam veteran PTSD patients treated with direct therapeutic exposure. Behavior Therapy. 1990;21 (1):63-87.
- [Background] Britt TW. The stigma of psychological problems in a work environment: Evidence from the screening of Service Members returning from Bosnia. J of Applied Psych. 2000;30(8):1599-1618
- [Background] Foa EB, Riggs DS, Massie ED, Yarczower M. The impact of fear activation and anger on the efficacy of exposure treatment for PTSD. Behavior Therapy. 1995;26:487-499.
- [Background] Rizzo AA, Buckwalter JG, van der Zaag C. Virtual Environment Applications for Neuropsychological Assessment and Rehabilitation. In: Stanney K, ed. Handbook of Virtual Environments. New York: L.A. Earlbaum; 2002:1027-1064.
- [Background] Smith SG, Rothbaum BO, Hodges L. Treatment of fear of flying using virtual reality exposure therapy: A single case study. The Behavior Therapist. 1999;22(8):154-158,160.
- [Background] Anderson P, Rothbaum BO, Hodges LF. Virtual reality exposure in the treatment of social anxiety: Two case reports. Cognitive and Behavioral Practice. 2003;10:240-247.
- [Background] Glantz K, Rizzo AA, Graap K. Virtual reality for psychotherapy: Current reality and future possibilities. Psychotherapy: Theory, Research, Practice, Training. 2003;40(1/2):55-67.
- [Background] Rizzo AA, Schultheis MT, Kerns K, Mateer C. Analysis of assets for virtual applications in neuropsychology. Neuropsychological Rehabilitation. 2004;14(1/2):207-239.
- [Background] Rizzo AA, Rothbaum BO, Graap K. Virtual Reality Applications for Combat-Related Posttraumatic Stress Disorder. In: Figley CR, Nash WP, eds. For Those Who Bore the Battle: Combat Stress Injury Theory, Research, and Management. New York: Taylor and Francis Books; 2006.
- [Background] Rothbaum BO, Ruef AM, Litz BT, Han H, Hodges L. Virtual reality exposure therapy of combat-related PTSD: A case study using psychophysiological indicators of outcome. Journal of Cognitive Psychotherapy. 2003;17(2):163-177.
- [Background] Cohen J. Statistical Power Analysis for the Behavioral Sciences. Hillsdale: Lawrence Earlbaum Associates; 1988.
- [Background] Cohen J, Cohen P. Applied Multiple Regression/Correlation Analysis for the Behavioral Sciences. Hillsdale: Lawrence Earlbaum; 1983.
- [Background] Foa EB, Hembree E, Rothbaum BO. Prolonged Exposure Therapy for PTSD: Emotional Processing of Traumatic Experiences. New York: Oxford University Press; 2007.
- [Background] Nishith P, Resick PA. Adherence and competence rating scales for prolonged exposure treatment: Unpublished Rating Scale, University of Missouri-St. Louis; 1994.
- [Background] Ajzen I. From intentions to actions: A theory of planned behavior. In: Kuhl J, Beckman, J, eds. Action-Control: From Cognition to Behavior. Heidelberg: Springer; 1985:11-39.
- [Background] Komiya N, Good GE, Sherrod NB. Emotional openness as a predictor of college students' attitudes toward seeking psychological help. J Counsel Psychol. 2000;47(1):138-143.
- [Background] Kennedy RS, Lane NE, Berbaum KS, Lilienthal MG. Simulator Sickness Questionnaire: An enhanced method for quantifying simulator sickness. International Journal of Aviation Psychology. 1993;3(3):203-220.
- [Result] Rothbaum BO, Hodges LF. The use of virtual reality exposure in the treatment of anxiety disorders. Behav Modif. 1999 Oct;23(4):507-25. doi: 10.1177/0145445599234001. PMID 10533438
- [Result] Pole N. The psychophysiology of posttraumatic stress disorder: a meta-analysis. Psychol Bull. 2007 Sep;133(5):725-46. doi: 10.1037/0033-2909.133.5.725. PMID 17723027
- [Result] Jaycox LH, Foa EB, Morral AR. Influence of emotional engagement and habituation on exposure therapy for PTSD. J Consult Clin Psychol. 1998 Feb;66(1):185-92. doi: 10.1037//0022-006x.66.1.185. PMID 9489273
- [Result] Difede J, Cukor J, Jayasinghe N, Patt I, Jedel S, Spielman L, Giosan C, Hoffman HG. Virtual reality exposure therapy for the treatment of posttraumatic stress disorder following September 11, 2001. J Clin Psychiatry. 2007 Nov;68(11):1639-47. PMID 18052556
- [Result] Hoge CW, Castro CA, Messer SC, McGurk D, Cotting DI, Koffman RL. Combat duty in Iraq and Afghanistan, mental health problems, and barriers to care. N Engl J Med. 2004 Jul 1;351(1):13-22. doi: 10.1056/NEJMoa040603. PMID 15229303
- [Result] Kessler RC, Sonnega A, Bromet E, Hughes M, Nelson CB. Posttraumatic stress disorder in the National Comorbidity Survey. Arch Gen Psychiatry. 1995 Dec;52(12):1048-60. doi: 10.1001/archpsyc.1995.03950240066012. PMID 7492257
- [Result] Simms LJ, Watson D, Doebbeling BN. Confirmatory factor analyses of posttraumatic stress symptoms in deployed and nondeployed veterans of the Gulf War. J Abnorm Psychol. 2002 Nov;111(4):637-47. doi: 10.1037//0021-843x.111.4.637. PMID 12428777
- [Result] Hoge CW, Auchterlonie JL, Milliken CS. Mental health problems, use of mental health services, and attrition from military service after returning from deployment to Iraq or Afghanistan. JAMA. 2006 Mar 1;295(9):1023-32. doi: 10.1001/jama.295.9.1023. PMID 16507803
- [Result] Seal KH, Bertenthal D, Miner CR, Sen S, Marmar C. Bringing the war back home: mental health disorders among 103,788 US veterans returning from Iraq and Afghanistan seen at Department of Veterans Affairs facilities. Arch Intern Med. 2007 Mar 12;167(5):476-82. doi: 10.1001/archinte.167.5.476. PMID 17353495

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Prolonged Exposure Therapy (PE) | Virtual Reality Exposure Therapy (VRET) | Waitlist
Started | 54 | 54 | 54
Completed | 32 | 30 | 47
Not Completed | 22 | 24 | 7

BASELINE CHARACTERISTICS:
Population: All participants randomized to a treatment arm included in baseline data analysis
Groups:
- Total: Total of all reporting groups
Arm/Group | Prolonged Exposure Therapy (PE) | Virtual Reality Exposure Therapy (VRET) | Waitlist | Total
Number analyzed (Participants) | 54 | 54 | 54 | 162
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 54 | 54 | 54 | 162
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 30.89 (7.09) | 29.52 (6.47) | 30.39 (6.45) | 30.27 (6.66)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 2 | 1 | 6
  Male | 51 | 52 | 53 | 156
Region of Enrollment [Number; unit: participants]
  United States | 54 | 54 | 54 | 162

OUTCOME MEASURES:

1. Primary Outcome: Clinician-Administered PTSD Scale (CAPS)
Description: The CAPS is a structured interview that assesses all Diagnostic and Statistical Manual of Mental Disorders (DSM-IV) PTSD criteria in terms of frequency and intensity. We used total scores as the primary outcome. Minimum possible score was 0, maximum possible score was 136. Higher scores indicated higher levels of symptoms.
Time Frame: Screening Visit (Day 1)
Population: Baseline scores on the CAPS-W (last week reference)
Measure: Mean (Standard Deviation); unit: units on scale
Arm/Group | Prolonged Exposure Therapy (PE) | Virtual Reality Exposure Therapy (VRET) | Waitlist
Number analyzed (Participants) | 54 | 54 | 54
units on scale | 78.28 (16.35) | 80.44 (16.23) | 78.89 (16.87)

2. Primary Outcome: Clinician-Administered PTSD Scale (CAPS)
Description: The CAPS is a structured interview that assesses all DSM-IV PTSD criteria in terms of frequency and intensity. Scores are computed for Intrusion, Avoidance and Hyperarousal symptom clusters, as well as a Total score.We used total scores as the primary outcome. Minimum possible score was 0, maximum possible score was 136. Higher scores indicated higher levels of symptoms.
Time Frame: 2.5 weeks (or after treatment session 5)
Population: Participants who provided data at mid treatment
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Prolonged Exposure Therapy (PE) | Virtual Reality Exposure Therapy (VRET) | Waitlist
Number analyzed (Participants) | 39 | 36 | 52
units on a scale | 65.03 (29.19) | 71.19 (23.27) | 74.73 (21.78)

3. Primary Outcome: Clinician-Administered PTSD Scale (CAPS)
Description: as for outcome 2
Time Frame: 5 weeks (or after treatment session 10)
Population: Participants who provided outcome data at post treatment
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Prolonged Exposure Therapy (PE) | Virtual Reality Exposure Therapy (VRET) | Waitlist
Number analyzed (Participants) | 32 | 30 | 47
units on a scale | 44.28 (33.73) | 57.07 (32.32) | 68.06 (24.27)
Statistical Analysis 1: Comparison: Prolonged Exposure Therapy (PE) vs Waitlist; Test type: Superiority or Other; Slope = -22.34, Standard Deviation 4.69
Statistical Analysis 2: Comparison: Virtual Reality Exposure Therapy (VRET) vs Waitlist; Test type: Superiority or Other; Slope = -13.30, Standard Error of Mean 4.77
Statistical Analysis 3: Comparison: Prolonged Exposure Therapy (PE) vs Virtual Reality Exposure Therapy (VRET); Test type: Superiority or Other; Slope = 9.04, Standard Error of Mean 5.11

4. Primary Outcome: Clinician-Administered PTSD Scale (CAPS)
Description: as for outcome 2
Time Frame: 12 week follow up
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Prolonged Exposure Therapy (PE) | Virtual Reality Exposure Therapy (VRET)
Number analyzed (Participants) | 27 | 26
units on a scale | 36.63 (31.80) | 55.88 (31.10)
Statistical Analysis 1: Comparison: Prolonged Exposure Therapy (PE) vs Virtual Reality Exposure Therapy (VRET); Test type: Superiority or Other; Slope = 15.07, Standard Deviation 6.03

5. Primary Outcome: Clinician-Administered PTSD Scale (CAPS)
Description: as for outcome 2
Time Frame: 26 Week follow up
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Prolonged Exposure Therapy (PE) | Virtual Reality Exposure Therapy (VRET)
Number analyzed (Participants) | 24 | 17
units on a scale | 38.33 (28.49) | 54.47 (28.62)
Statistical Analysis 1: Comparison: Prolonged Exposure Therapy (PE) vs Virtual Reality Exposure Therapy (VRET); Test type: Superiority or Other; Slope = 13.91, Standard Error of Mean 6.70

6. Secondary Outcome: PTSD Checklist- Civilian (PCL-C)
Description: The PCL-C is a self report measure that evaluates att 17 PTSD criteria using a 5 point Likert scale.
Time Frame: Screening Visit (Day 1)
Reporting Status: Not Posted

7. Secondary Outcome: Primary Care PTSD Screen (PC-PTSD)
Description: The PC-PTSD is a four-item measure designed to screen for PTSD.
Time Frame: Screening Visit (Day 1)
Reporting Status: Not Posted

8. Secondary Outcome: Beck Depression Inventory-II (BDI-II)
Description: This self report measure of depression contains 21 items that are rated on a 4 point scale.
Time Frame: Screening Visit(Day 1)
Reporting Status: Not Posted

9. Secondary Outcome: Inventory of Attitudes Toward Seeking Mental Health Services (IASMHS)
Description: The IASMHS is a 24 item assessment of help-seeking attitudes. It includes the following three factors based on components of Ajzen's Theory of Planned Behavior: Psychological Openness, Help-seeking Propensity and Indifference to Stigma.
Time Frame: Screening Visit(Day 1)
Reporting Status: Not Posted

10. Secondary Outcome: Perceived Stigma Measure (PSS)
Description: Stigma will be measured using a 5 question assessment scale.
Time Frame: Screening Visit(Day 1)
Reporting Status: Not Posted

11. Secondary Outcome: Suicide Risk Assessment
Description: Due to the nature of the questions, this is deemed to be of safety nature.
Time Frame: Screening Visit(Day 1)
Reporting Status: Not Posted

12. Secondary Outcome: Beck Anxiety Inventory (BAI)
Description: The BAI is a self report measure consisting of 21 items designed to discriminate anxiety from depression.
Time Frame: Screening Visit(Day 1)
Reporting Status: Not Posted

13. Secondary Outcome: Behavior and Sympton Identification Scale (BASIS-24)
Description: To assess overall psychological pain and gives an indicator of overall wellness. Due to the nature of the questions, this is deemed to be of safety nature.
Time Frame: Screening Visit(Day 1)
Reporting Status: Not Posted

14. Secondary Outcome: Intent to Attend
Description: This is a measure to assess the intent to complete study procedures.
Time Frame: Screening Visit (Day 1)
Reporting Status: Not Posted

15. Secondary Outcome: Subjective Units of Distress (SUDs)
Description: Ranging from 1 to 100, Subjective Units of Distress are gathered every 5 mintues during imaginal exposure to determine levels of distress and engagement in the situation.
Time Frame: Treatment session 1 (week 1)
Reporting Status: Not Posted

16. Secondary Outcome: Side Effects Questionnaire
Description: The Side Effects Questionnaire is based on a revised version of the Simulator Sickness Questionnaire (SSQ) that will be used to measure general discomfort in both the VRET and PE conditions of the study.
Time Frame: Treatment session 1(week 1)
Reporting Status: Not Posted

17. Secondary Outcome: BASIS-24
Description: as for outcome 13
Time Frame: Treatment session 1 (week 1)
Reporting Status: Not Posted

18. Secondary Outcome: Intent to Attend
Description: This is a measure to assess the intent to complete study procedures.
Time Frame: Treatment session 1 (week 1)
Reporting Status: Not Posted

19. Secondary Outcome: PTSD Checklist (PCL-C)
Description: The PCL-C is a self report measure that evaluates att 17 PTSD criteria using a 5 point Likert scale.
Time Frame: 2.5 weeks (or after treatment session 5)
Reporting Status: Not Posted

20. Secondary Outcome: PTSD Checklist (PCL-C)
Description: The PCL-C is a self report measure that evaluates att 17 PTSD criteria using a 5 point Likert scale.
Time Frame: 5 weeks (or after treatment session 10)
Reporting Status: Not Posted

21. Secondary Outcome: Primary Care PTSD Screen (PC-PTSD)
Description: The PC-PTSD is a four-item measure designed to screen for PTSD.
Time Frame: 2.5 weeks (or after treatment session 5)
Reporting Status: Not Posted

22. Secondary Outcome: PTSD Checklist (PCL-C)
Description: The PCL-C is a self report measure that evaluates att 17 PTSD criteria using a 5 point Likert scale.
Time Frame: 12 week follow up
Reporting Status: Not Posted

23. Secondary Outcome: PTSD Checklist (PCL-C)
Description: The PCL-C is a self report measure that evaluates att 17 PTSD criteria using a 5 point Likert scale.
Time Frame: 26 week follow up
Reporting Status: Not Posted

24. Secondary Outcome: Primary Care PTSD Screen (PC-PTSD)
Description: The PC-PTSD is a four-item measure designed to screen for PTSD.
Time Frame: 5 weeks (or after treatment session 10)
Reporting Status: Not Posted

25. Secondary Outcome: Primary Care PTSD Screen (PC-PTSD)
Description: The PC-PTSD is a four-item measure designed to screen for PTSD.
Time Frame: 12 Week follow up
Reporting Status: Not Posted

26. Secondary Outcome: Primary Care PTSD Screen (PC-PTSD)
Description: The PC-PTSD is a four-item measure designed to screen for PTSD.
Time Frame: 26 Week follow up
Reporting Status: Not Posted

27. Secondary Outcome: Beck Depression Inventory-II (BDI-II)
Description: This self report measure of depression contains 21 items that are rated on a 4 point scale.
Time Frame: 2.5 weeks (or after treatment session 5)
Reporting Status: Not Posted

28. Secondary Outcome: Beck Depression Inventory-II (BDI-II)
Description: This self report measure of depression contains 21 items that are rated on a 4 point scale.
Time Frame: 5 weeks (or after treatment session 10)
Reporting Status: Not Posted

29. Secondary Outcome: Beck Depression Inventory-II (BDI-II)
Description: This self report measure of depression contains 21 items that are rated on a 4 point scale.
Time Frame: 12 Week follow up
Reporting Status: Not Posted

30. Secondary Outcome: Beck Depression Inventory-II (BDI-II)
Description: This self report measure of depression contains 21 items that are rated on a 4 point scale.
Time Frame: 26 Week follow up
Reporting Status: Not Posted

31. Secondary Outcome: Inventory of Attitudes Toward Seeking Mental Health Services (IASMHS)
Description: as for outcome 9
Time Frame: 2.5 weeks (or after treatment session 5)
Reporting Status: Not Posted

32. Secondary Outcome: Inventory of Attitudes Toward Seeking Mental Health Services (IASMHS)
Description: as for outcome 9
Time Frame: 5 weeks (or after treatment session 10)
Reporting Status: Not Posted

33. Secondary Outcome: Inventory of Attitudes Toward Seeking Mental Health Services (IASMHS)
Description: as for outcome 9
Time Frame: 12 Week follow up
Reporting Status: Not Posted

34. Secondary Outcome: Inventory of Attitudes Toward Seeking Mental Health Services (IASMHS)
Description: as for outcome 9
Time Frame: 26 Week follow up
Reporting Status: Not Posted

35. Secondary Outcome: Perceived Stigma Measure (PSS)
Description: Stigma will be measured using a 5 question assessment scale.
Time Frame: 2.5 weeks (or after treatment session 5)
Reporting Status: Not Posted

36. Secondary Outcome: Perceived Stigma Measure (PSS)
Description: Stigma will be measured using a 5 question assessment scale.
Time Frame: 5 weeks (or after treatment session 10)
Reporting Status: Not Posted

37. Secondary Outcome: Perceived Stigma Measure (PSS)
Description: Stigma will be measured using a 5 question assessment scale.
Time Frame: 12 week follow up
Reporting Status: Not Posted

38. Secondary Outcome: Perceived Stigma Measure (PSS)
Description: Stigma will be measured using a 5 question assessment scale.
Time Frame: 26 week follow up
Reporting Status: Not Posted

39. Secondary Outcome: Suicide Risk Assessment
Description: Due to the nature of the questions, this is deemed to be of safety nature.
Time Frame: 2.5 weeks (or after treatment session 5)
Reporting Status: Not Posted

40. Secondary Outcome: Suicide Risk Assessment
Description: Due to the nature of the questions, this is deemed to be of safety nature.
Time Frame: 5 weeks (or after treatment session 10)
Reporting Status: Not Posted

41. Secondary Outcome: Suicide Risk Assessment
Description: Due to the nature of the questions, this is deemed to be of safety nature.
Time Frame: 12 Week follow up
Reporting Status: Not Posted

42. Secondary Outcome: Suicide Risk Assessment
Description: Due to the nature of the questions, this is deemed to be of safety nature.
Time Frame: 26 Week follow up
Reporting Status: Not Posted

43. Secondary Outcome: Beck Anxiety Inventory (BAI)
Description: The BAI is a self report measure consisting of 21 items designed to discriminate anxiety from depression.
Time Frame: 2.5 weeks (or after treatment session 5)
Reporting Status: Not Posted

44. Secondary Outcome: Beck Anxiety Inventory (BAI)
Description: The BAI is a self report measure consisting of 21 items designed to discriminate anxiety from depression.
Time Frame: 5 weeks (or after treatment session 10)
Reporting Status: Not Posted

45. Secondary Outcome: Beck Anxiety Inventory (BAI)
Description: The BAI is a self report measure consisting of 21 items designed to discriminate anxiety from depression.
Time Frame: 12 week follow up
Reporting Status: Not Posted

46. Secondary Outcome: Beck Anxiety Inventory (BAI)
Description: The BAI is a self report measure consisting of 21 items designed to discriminate anxiety from depression.
Time Frame: 26 week follow up
Reporting Status: Not Posted

47. Secondary Outcome: BASIS-24
Description: as for outcome 13
Time Frame: Treatment session 2 (week 1)
Reporting Status: Not Posted

48. Secondary Outcome: BASIS-24
Description: as for outcome 13
Time Frame: Treatment session 3 (week 2)
Reporting Status: Not Posted

49. Secondary Outcome: BASIS-24
Description: as for outcome 13
Time Frame: Treatment session 4 (week 2)
Reporting Status: Not Posted

50. Secondary Outcome: BASIS-24
Description: as for outcome 13
Time Frame: Treatment session 5 (week 2.5)
Reporting Status: Not Posted

51. Secondary Outcome: BASIS-24
Description: as for outcome 13
Time Frame: Treatment session 6 (week 3)
Reporting Status: Not Posted

52. Secondary Outcome: BASIS-24
Description: as for outcome 13
Time Frame: Treatment session 7 (week 4)
Reporting Status: Not Posted

53. Secondary Outcome: BASIS-24
Description: as for outcome 13
Time Frame: Treatment session 8 (week 4)
Reporting Status: Not Posted

54. Secondary Outcome: BASIS-24
Description: as for outcome 13
Time Frame: Treatment session 9 (week 5)
Reporting Status: Not Posted

55. Secondary Outcome: BASIS-24
Description: as for outcome 13
Time Frame: Treatment session 10 (week 5)
Reporting Status: Not Posted

56. Secondary Outcome: BASIS-24
Description: as for outcome 13
Time Frame: 5 weeks (or after treatment session 10)
Reporting Status: Not Posted

57. Secondary Outcome: BASIS-24
Description: as for outcome 13
Time Frame: 2.5 weeks (or after treatment session 5)
Reporting Status: Not Posted

58. Secondary Outcome: BASIS-24
Description: as for outcome 13
Time Frame: 12 week follow up
Reporting Status: Not Posted

59. Secondary Outcome: BASIS-24
Description: as for outcome 13
Time Frame: 26 week follow up
Reporting Status: Not Posted

60. Secondary Outcome: Subjective Units of Distress (SUDs)
Description: as for outcome 15
Time Frame: Treatment session 2 (week 1)
Reporting Status: Not Posted

61. Secondary Outcome: Subjective Units of Distress (SUDs)
Description: as for outcome 15
Time Frame: Treatment session 3 (week 2)
Reporting Status: Not Posted

62. Secondary Outcome: Subjective Units of Distress (SUDs)
Description: as for outcome 15
Time Frame: Treatment session 4 (week 2)
Reporting Status: Not Posted

63. Secondary Outcome: Subjective Units of Distress (SUDs)
Description: as for outcome 15
Time Frame: Treatment session 5 (week 2.5)
Reporting Status: Not Posted

64. Secondary Outcome: Subjective Units of Distress (SUDs)
Description: as for outcome 15
Time Frame: Treatment session 6 (week 3)
Reporting Status: Not Posted

65. Secondary Outcome: Subjective Units of Distress (SUDs)
Description: as for outcome 15
Time Frame: Treatment session 7 (week 4)
Reporting Status: Not Posted

66. Secondary Outcome: Subjective Units of Distress (SUDs)
Description: as for outcome 15
Time Frame: Treatment session 8 (week 4)
Reporting Status: Not Posted

67. Secondary Outcome: Subjective Units of Distress (SUDs)
Description: as for outcome 15
Time Frame: Treatment session 9 (week 5)
Reporting Status: Not Posted

68. Secondary Outcome: Subjective Units of Distress (SUDs)
Description: as for outcome 15
Time Frame: Treatment session 10 (week 5)
Reporting Status: Not Posted

69. Secondary Outcome: Side Effects Questionnaire
Description: as for outcome 16
Time Frame: Treatment session 2 (week 1)
Reporting Status: Not Posted

70. Secondary Outcome: Side Effects Questionnaire
Description: as for outcome 16
Time Frame: Treatment session 3 (week 2)
Reporting Status: Not Posted

71. Secondary Outcome: Side Effects Questionnaire
Description: as for outcome 16
Time Frame: Treatment session 4 (week 2)
Reporting Status: Not Posted

72. Secondary Outcome: Side Effects Questionnaire
Description: as for outcome 16
Time Frame: Treatment session 5 (week 2.5)
Reporting Status: Not Posted

73. Secondary Outcome: Side Effects Questionnaire
Description: as for outcome 16
Time Frame: Treatment session 6 (week 3)
Reporting Status: Not Posted

74. Secondary Outcome: Side Effects Questionnaire
Description: as for outcome 16
Time Frame: Treatment session 7 (week 4)
Reporting Status: Not Posted

75. Secondary Outcome: Side Effects Questionnaire
Description: as for outcome 16
Time Frame: Treatment session 8 (week 4)
Reporting Status: Not Posted

76. Secondary Outcome: Side Effects Questionnaire
Description: as for outcome 16
Time Frame: Treatment session 9 (week 5)
Reporting Status: Not Posted

77. Secondary Outcome: Side Effects Questionnaire
Description: as for outcome 16
Time Frame: Treatment session 10 (week 5)
Reporting Status: Not Posted

78. Secondary Outcome: Intent to Attend
Description: This is a measure to assess the intent to complete study procedures.
Time Frame: Treatment session 2 (week 1)
Reporting Status: Not Posted

79. Secondary Outcome: Intent to Attend
Description: This is a measure to assess the intent to complete study procedures.
Time Frame: Treatment session 3 (week 2)
Reporting Status: Not Posted

80. Secondary Outcome: Intent to Attend
Description: This is a measure to assess the intent to complete study procedures.
Time Frame: Treatment session 4 (week 2)
Reporting Status: Not Posted

81. Secondary Outcome: Intent to Attend
Description: This is a measure to assess the intent to complete study procedures.
Time Frame: Treatment session 5 (week 2.5)
Reporting Status: Not Posted

82. Secondary Outcome: Intent to Attend
Description: This is a measure to assess the intent to complete study procedures.
Time Frame: Treatment session 6 (week 3)
Reporting Status: Not Posted

83. Secondary Outcome: Intent to Attend
Description: This is a measure to assess the intent to complete study procedures.
Time Frame: Treatment session 7 (week 4)
Reporting Status: Not Posted

84. Secondary Outcome: Intent to Attend
Description: This is a measure to assess the intent to complete study procedures.
Time Frame: Treatment session 8 (week 4)
Reporting Status: Not Posted

85. Secondary Outcome: Intent to Attend
Description: This is a measure to assess the intent to complete study procedures.
Time Frame: Treatment session 9 (week 5)
Reporting Status: Not Posted

86. Secondary Outcome: Intent to Attend
Description: This is a measure to assess the intent to complete study procedures.
Time Frame: Treatment session 10 (week 5)
Reporting Status: Not Posted

87. Secondary Outcome: Intent to Attend
Description: This is a measure to assess the intent to complete study procedures.
Time Frame: 2.5 weeks (or after treatment session 5)
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 6 months. From time of baseline visit to final follow up visit
Arm/Group | Prolonged Exposure Therapy (PE) | Virtual Reality Exposure Therapy (VRET) | Waitlist
Serious Adverse Events (participants affected / at risk) | 0/54 | 3/54 | 0/54
Other Adverse Events (participants affected / at risk) | 12/54 | 15/54 | 0/54
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Prolonged Exposure Therapy (PE) (N=54) | Virtual Reality Exposure Therapy (VRET) (N=54) | Waitlist (N=54)
Hospitalization - psychiatric (Psychiatric disorders) | 0 (0) | 3 (3) | 0 (0) — All three SAE's were for psychiatric hospitalization - not related to study
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Prolonged Exposure Therapy (PE) (N=54) | Virtual Reality Exposure Therapy (VRET) (N=54) | Waitlist (N=54)
increase in flashbacks (Psychiatric disorders) | 1 (3) | 0 (0) | 0 (0)
Headache (General disorders) | 7 (9) | 4 (8) | 0 (0) — Headaches
Dislocated Shoulder (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) — Shoulder dislocation during racket ball which was in in vivo homework exercise
exacerbation of neck and back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2) | 0 (0)
chest pain (Cardiac disorders) | 1 (1) | 1 (2) | 0 (0)
Nausea (Gastrointestinal disorders) | 5 (6) | 3 (4) | 0 (0)
Eczema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (2) | 0 (0)
dizziness (General disorders) | 2 (2) | 1 (1) | 0 (0)
homicidal ideation (Psychiatric disorders) | 0 (0) | 2 (2) | 0 (0)
intermittent stomach ache and diarrhea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
increased intrusive memories (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
increased irritability (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Shortness of Breath (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
increased anxiety around weapons (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
flu like symptoms (General disorders) | 0 (0) | 1 (2) | 0 (0)
cold symptoms (General disorders) | 0 (0) | 1 (1) | 0 (0)
syncopal episode (General disorders) | 1 (1) | 0 (0) | 0 (0)
rash from ECG lead (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
alcohol consumption (General disorders) | 2 (2) | 0 (0) | 0 (0) — Alcohol consumption after session
self percieved persecution (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) — starving self, vague suicidal ideation and homicidal ideation

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No